CLINICAL TRIAL: NCT06781749
Title: New Approach to Objectively Measure Social Engagement in Older Adults With Hearing Loss
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Janet Choi, Assistant Professor, University of Southern California
Other Study IDs: UP-24-01177
Record Dates: First submitted 2025-01-08; First posted 2025-01-17 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Hearing Loss, Bilateral (Causes Other Than Tumors)
Keywords: hearing loss; hearing aids; cognition; dementia
MeSH Terms: conditions — Hearing Loss; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adults with bilateral hearing loss (hearing aid users): Participants with bilateral hearing loss (defined as those with speech-frequency pure-tone average >=25 dB HL bilaterally) and currently using hearing aids.
  Interventions: Device: Hearing aid use
- Adults without hearing loss: Hearing loss defined as speech-frequency pure-tone average >=25 dB HL bilaterally
- Adults with hearing loss (non-hearing aid users): Participants with bilateral hearing loss (defined as those with speech-frequency pure-tone average >=25 dB HL bilaterally) and not currently using hearing aids.

INTERVENTIONS:
Device: Hearing aid use — Hearing aid use will be discussed with all eligible participants with hearing loss and will be encouraged to pursue hearing aid fitting through standard clinical indications via participants' insurance and audiologists.
  Groups: Adults with bilateral hearing loss (hearing aid users)

SUMMARY:
The goal of this clinical trial is to learn if hearing devices, like hearing aids, affect social and cognitive function of older adults. The main questions the researchers want to answer are:

* How social are older adults with hearing loss before and after using hearing devices?
* How well do older adults with hearing loss think before and after using hearing devices?
* For older adults who have hearing loss and use hearing devices, do changes in social interaction explain changes in how well they think (cognitive function)?
* Do brainwaves (EEGs) in older adults with hearing loss change after using hearing devices?
* Are there differences in how social older adults with hearing loss are compared to older adults without hearing loss?

What Participants Will Do:

* Participants will take questionnaires for around 60 minutes. Questionnaires will ask participants about their background, health, hearing, and how social they are. Another set of questionnaires will check their thinking ability or cognition.
* Participants will wear an audio sensor (TILES Audio Recorder on Jelly Mobile phone) for 2 weeks. The sensor will collect and store information about a participant's voice during conversations. Once the device has information about a participant's voice such as pitch and tone it will store this information and delete the audio recording. Words spoken during conversations will be deleted.
* (Optional) Participants can choose to participate in a 45-60-minute EEG (electroencephalogram) recording session. Participants will have sensors placed on top of their heads. Sensors will record the participants' brainwaves. Sounds will be played to see how participants' brainwaves change when they hear sounds. Eligible participants will be invited to participate in 4-month follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 60 years
* English or Spanish speaking
* Group 1- older adults with normal hearing defined as speech frequency PTA <25dB HL in bilateral ears
* Group 2- older adults with bilateral hearing loss who are not using hearing aids
* Group 3- older adults with bilateral hearing loss, who are currently using hearing aids

Exclusion Criteria:

* Age <60 years
* Unable to complete questionnaires in English or Spanish

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals meeting the inclusion criteria will be recruited from the affiliated tertiary hospitals and hearing aid centers. Both individuals with audiometry-measured bilateral hearing loss who are clinically indicated for hearing aid fitting and healthy volunteers without hearing loss will be recruited to participant in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive test- MoCA | Baseline and 4-month after hearing aid use
  MoCA (MoCA-Basic if appropriate) score

SECONDARY OUTCOMES:
Cognitive Test- Digit Span Test | Baseline, 4-month after hearing aid use
  Cognitive Test- Digit Span Test
Audio sensor- speech arousal | Baseline, 4-month after hearing aid use
  The audio sensor employs deep-learning-based multimodal speech pattern modeling of participants' own voice activities to extract speech arousal and speech activities. Speech arousal measures include the percentage of strong arousals, serving as a proxy of enhanced engagement in conversations.
Audio sensor- speech activity | Baseline and 4-month after hearing aid use
  The audio sensor employs deep-learning-based multimodal speech pattern modeling of participants' own voice activities to extract speech arousal and speech activities. Speech activity measures include the intersession time (the interval between speech sessions, representing the frequency of conversation engagement).
EEG Measures | Baseline, 4-month after hearing aid use
  EEG Event Related Potentials (ERPs) are measures of cortical activities in response to auditory stimuli and provide information about cognitive processing, memory, and attention. Participants will complete auditory oddball tasks during EEG measurements and ERPs including P1, N1, P2, MMN, P3 will be recorded.
Auditory oddball task | Baseline and 4-mo after hearing aid use
  Auditory oddball task discrimination sensitivity

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Los Angeles General Medical Center, Los Angeles, California
  - University of Southern California, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No